CLINICAL TRIAL: NCT01537133
Title: Airway Microbiome in Asthma: Relationships to Asthma Phenotype and Inhaled Corticosteroid Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Professor of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: AsthmaNet 003; U10HL098115 (NIH)
Record Dates: First submitted 2012-02-09; First posted 2012-02-23 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Asthma; Atopy
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Inhaled corticosteroid (Experimental): Fluticasone (250 mcg/puff, one puff, twice a day)
  Interventions: Drug: fluticasone
- Placebo (Placebo Comparator): Placebo fluticasone (one puff, twice a day)
  Interventions: Drug: Placebo
- Healthy Control (No Intervention)
- Atopic Non-asthmatics (No Intervention)

INTERVENTIONS:
Drug: fluticasone — Dry Powder Inhaler: 250 mcg/puff, one puff, twice a day
  Other Names: Flovent 250
  Arms: Inhaled corticosteroid
Drug: Placebo — Dry Powder Inhaler: Placebo
  Arms: Placebo

SUMMARY:
There are new, very sensitive methods for detecting bacteria. These methods show that hundreds of millions of microbes (organisms that can only be seen with microscopes), especially bacteria, live in healthy people. The collection of different microbes found in a site is called a "microbiome." The investigators know that microbiomes of the skin, sinuses, mouth, gastro-intestinal tract, etc. differ from each other. The make-up of the microbiome - which bacteria are found in a site - may be necessary for good health. For example, the microbiome of the mouth is different in people with inflammation of the gums (periodontitis), and the microbiome of the bowel is different in people with inflammation of the intestinal tract (inflammatory bowel disease).

The purpose of this research study is to find out if the microbiome in the lungs is different in healthy people without asthma compared to people with asthma. This study will also find out if the microbiome of the lungs changes when people with asthma take a daily "controller" medication called an inhaled corticosteroid.

DETAILED DESCRIPTION:
Two broad specific aims of this study are: 1)To evaluate whether the microbiota of the bronchial airways in atopic asthmatics and atopic healthy controls differ in microbial diversity, richness, evenness, or composition of specific bacterial taxa. 2) To determine whether inhaled corticosteroid treatment alters bronchial microbial community composition in asthmatics.

ELIGIBILITY:
Inclusion Criteria:

Asthmatic:

* History of physician-diagnosed asthma.
* Methacholine PC20 < 8mg/ml and/or FEV1 improvement ≥ 12% in response to 180 mcg albuterol.
* FEV1 ≥ 70% of predicted after 180 mcg albuterol.
* Stable asthma for ≥ 3 months prior to enrollment (no urgent care visits, no systemic corticosteroid treatment).
* Asthma Control Questionnaire 6 Score < 1.5.
* Able to provide informed consent.
* Able to perform spirometry as per ATS criteria.
* Evidence by allergen skin test of sensitivity to an aeroallergen.
* Willingness, if female and able to conceive, to utilize one medically-acceptable form of contraception.

Healthy Control:

* Evidence by allergen skin test of sensitivity to an aeroallergen.
* Able to provide informed consent.
* Able to perform spirometry as per ATS criteria.

Exclusion Criteria:

Asthmatic:

* Presence of lung disease other than asthma.
* Use of > 10 doses of nasal corticosteroids in the previous 3 months.
* Presence of significant medical illness or other chronic diseases whose treatment could affect the clinical features measured, responses to the therapies to be given in this study, or risks of participating in the study.
* History of atrial or ventricular tachyarrhythmia.
* Changes suggestive of cardiac ischemia on ECG at baseline.
* History of upper respiratory infection, sinusitis, bronchitis, or antibiotic use in the previous 3 months.
* History of chronic sinus disease.
* Smoking > 5 pack-years, or within the past year
* History of long-term controller medication use for asthma (inhaled or oral corticosteroid, leukotriene pathway antagonist, cromolyn, or theophylline within the preceding 6 months.
* History of bleeding disorder.
* Reduced creatinine clearance.
* Inability, in the opinion of the Study Investigator, to coordinate use of inhaler or otherwise comply with medication regimens.
* Contraindication to bronchoscopy on history or examination.

Healthy Control:

* History of chronic respiratory disease including asthma.
* Presence of significant medical illness or other chronic diseases whose treatment could affect the clinical features measured, responses to the therapies to be given in this study, or risks of participating in the study.
* History of atrial or ventricular tachyarrhythmia.
* Changes suggestive of cardiac ischemia on ECG at baseline.
* History of upper respiratory infection, sinusitis, bronchitis, or antibiotic use in the previous 3 months.
* Methacholine PC20 < 16 mg/ml or FEV1 improvement ≥ 12% in response to albuterol.
* History of chronic sinus disease
* Smoking > 5 pack-years, or within the past year
* Use of > 10 doses of a nasal corticosteroid preparation in the previous 3 months
* FEV1 or FVC < 80% predicted.
* History of bleeding disorder.
* Reduced creatinine clearance.
* Contraindication to bronchoscopy on history or examination.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Lewis Smith, MD, Principal Investigator — Northwestern Memorial Hospital; Richard Martin, MD, Principal Investigator — National Jewish Health; Mario Castro, MD, Principal Investigator — Washington University School of Medicine; Monica Kraft, MD, Principal Investigator — Duke University; Stephen Peters, MD, Principal Investigator — Wake Forest University Health Sciences; Homer Boushey, MD, Principal Investigator — University of California, San Francisco; Sally Wenzel, MD, Principal Investigator — University of Pittsburgh Medical Center; Christine Sorkness, MD, Principal Investigator — University of Wisconsin, Madison
Locations (9):
- United States (9):
  - University of California, San Francisco, Adult, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University School of Medicine, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Pittsburgh, Adult, Pittsburgh, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Durack J, Christian LS, Nariya S, Gonzalez J, Bhakta NR, Ansel KM, Beigelman A, Castro M, Dyer AM, Israel E, Kraft M, Martin RJ, Mauger DT, Peters SP, Rosenberg SR, Sorkness CA, Wechsler ME, Wenzel SE, White SR, Lynch SV, Boushey HA, Huang YJ; National Heart, Lung, and Blood Institute's "AsthmaNet". Distinct associations of sputum and oral microbiota with atopic, immunologic, and clinical features in mild asthma. J Allergy Clin Immunol. 2020 Nov;146(5):1016-1026. doi: 10.1016/j.jaci.2020.03.028. Epub 2020 Apr 13. PMID 32298699

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy controls and non-atopic asthmatics assessed only at baseline.
Period: Overall Study
Arm/Group | Inhaled Corticosteroid | Placebo | Healthy Control | Atopic Non-asthmatics
Started | 28 | 14 | 21 | 21
Completed | 25 | 14 | 21 | 21
Not Completed | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atopic Asthmatics Treated With Inhaled Corticosteroid: Fluticasone (250 mcg/puff, one puff, twice a day)
- Atopic Asthmatics Treated With Placebo: Placebo fluticasone (one puff, twice a day)
- Total: Total of all reporting groups
Arm/Group | Atopic Asthmatics Treated With Inhaled Corticosteroid | Atopic Asthmatics Treated With Placebo | Atopic Non-asthmatics | Healthy Control | Total
Number analyzed (Participants) | 28 | 14 | 21 | 21 | 84
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [26 to 40] | 37 [25 to 40] | 28 [25 to 42] | 28 [24 to 45] | 30 [25 to 42]
Gender [Count of Participants; unit: Participants]
  Female | 16 | 7 | 11 | 12 | 46
  Male | 12 | 7 | 10 | 9 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16 | 9 | 11 | 15 | 51
  Black | 7 | 3 | 6 | 3 | 19
  Hispanic or Latio | 3 | 0 | 0 | 2 | 5
  Other | 2 | 2 | 4 | 1 | 9
Forced Expiratory Volume in 1 second [Median (Inter-Quartile Range); unit: percent of predicted] | 94 [76 to 99] | 84 [77 to 89] | 98 [89 to 108] | 100 [94 to 107] | 96 [86 to 105]
Blood Eosinophils [Median (Inter-Quartile Range); unit: percent of cells in blood sample] | 3.3 [1.3 to 5.7] | 3.6 [2 to 4.8] | 2.0 [1.4 to 2.9] | 1.4 [1.0 to 3.0] | 2.0 [1.2 to 4.0]
Sputum eosinophils [Median (Inter-Quartile Range); unit: percent of cells in sputum sample] | 0.3 [0.0 to 0.8] | 0.7 [0 to 1.5] | 0 [0 to 0.45] | 0 [0 to 0.4] | 0.2 [0.0 to 0.6]

OUTCOME MEASURES:

1. Primary Outcome: Microbial Community Richness
Description: Richness is the total number of different bacterial taxa detected in the sample.
Time Frame: baseline and after 6 weeks of treatment
Population: Only baseline samples were collected from atopic non-asthmatics and healthy controls. Data was not available for all participants due to insufficient amplification in some samples.
Measure: Median (Inter-Quartile Range); unit: number of bacterial taxa
Arm/Group | Atopic Asthmatics Treated With Inhaled Corticosteroids | Atopic Asthmatics Treated With Placebo | Atopic Non-asthmatics | Healthy Control
Number analyzed (Participants) | 16 | 12 | 15 | 13
number of bacterial taxa
  baseline | 449 [376 to 613] | 543 [484 to 684] | 483 [437 to 646] | 444 [400 to 530]
  after 6 weeks of treatment | 456 [351 to 578] | 405 [385 to 714] | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls

2. Primary Outcome: Microbial Community Diversity
Description: The Shannon diversity index is a type of entropy measure and is a function of the distribution of the total number of organisms across all of the species. If S is the total number of species in the sample and p_i is the number of organisms in the i-th species divided by the total number of organisms, then Diversity = -Σ p_i log(p_i).
Time Frame: baseline and after 6 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Shannon Diversity Index
Arm/Group | Atopic Asthmatics Treated With Inhaled Corticosteroids | Atopic Asthmatics Treated With Placebo | Atopic Non-asthmatics | Healthy Control
Number analyzed (Participants) | 16 | 12 | 15 | 13
Shannon Diversity Index
  baseline | 5.4 [4.9 to 5.6] | 5.7 [5.0 to 6.0] | 5.6 [5.2 to 6.0] | 5.3 [5.2 to 5.5]
  after 6 weeks of treatment | 5.0 [4.6 to 5.7] | 5.1 [4.8 to 5.7] | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls

3. Primary Outcome: Microbial Community Evenness
Description: Pielou's evenness index is a scaled measure of biodiversity and is equal to the observed Shannon diversity index divided by the maximum possible Shannon diversity index, which would occur if all of the species in the sample were equally abundant. Evenness = D/log(S), where D is the Shannon Diversity index and log(S) is the maximum diversity of the sample.
Time Frame: baseline and after 6 weeks of treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Pielou's evenness index
Arm/Group | Atopic Asthmatics Treated With Inhaled Corticosteroids | Atopic Asthmatics Treated With Placebo | Atopic Non-asthmatics | Healthy Control
Number analyzed (Participants) | 16 | 12 | 15 | 13
Pielou's evenness index
  baseline | 0.88 [0.81 to 0.90] | 0.88 [0.79 to 0.91] | 0.90 [0.83 to 0.94] | 0.86 [0.83 to 0.91]
  after 6 weeks of treatment | 0.85 [0.76 to 0.90] | 0.86 [0.81 to 0.88] | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls | NA [NA to NA] — Only baseline data was collected from atopic non-asthmatics and healthy controls

ADVERSE EVENTS:
Description: Adverse events were not collected or assessed for healthy controls or atopic non-asthmatics
Arm/Group | Inhaled Corticosteroid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/14
Other Adverse Events (participants affected / at risk) | 2/28 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Corticosteroid (N=28) | Placebo (N=14)
Acute nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No